CLINICAL TRIAL: NCT01471782
Title: A Single-Arm Multicenter Phase II Study Preceded by Dose Evaluation to Investigate the Efficacy, Safety, and Tolerability of the BiTE® Antibody Blinatumomab (MT103) in Pediatric and Adolescent Patients With Relapsed/Refractory B-Precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Clinical Study With Blinatumomab in Pediatric and Adolescent Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT103-205; 2010-024264-18 (EudraCT Number)
Record Dates: First submitted 2011-10-28; First posted 2011-11-16 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; relapsed, refractory B-precursor ALL; Leukemia; Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Antibodies, Bispecific
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Burkitt Lymphoma; Leukemia; Leukemia, Lymphoid; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): Blinatumomab was administered as a continuous intravenous (cIV) infusion at a constant daily flow rate over 4 weeks followed by a treatment-free interval of 2 weeks. Doses ranged between 5 and 30 µg/m²/day. Each participant received up to five cycles of treatment.
  Interventions: Biological: Blinatumomab

INTERVENTIONS:
Biological: Blinatumomab — Administered by continuous intravenous infusion
  Other Names: MT103; AMG103; BLINCYTO®

SUMMARY:
The purpose of this study is to determine the dose of the bispecific T cell engager blinatumomab (MT103) in pediatric and adolescent patients with relapsed/refractory acute lymphoblastic leukemia (ALL) and to assess whether this dose of blinatumomab is effective.

DETAILED DESCRIPTION:
Childhood acute lymphoblastic leukemia (ALL) is a type of cancer of the blood and bone marrow in which the bone marrow makes too many abnormal immature lymphocytes.

Blinatumomab is a bispecific single-chain antibody construct designed to link B cells and T cells resulting in T cell activation and a cytotoxic T cell response against cluster of differentiation (CD)19 expressing cells.

The purpose of this study is to investigate the pharmacokinetics (PK), pharmacodynamics (PD) and safety of escalating doses of blinatumomab in pediatric and adolescent patients with relapsed/refractory B-precursor ALL, to select a dose and to investigate the efficacy and safety of that dose of blinatumomab in the above-mentioned patient population.

The phase 1 part of the study included the evaluation of four dose levels of blinatumomab with comprehensive PK/PD assessments and was separated in 2 parts:

* Phase 1 dose evaluation/escalation part to define the recommended phase 2 dose of blinatumomab in patients aged 2 to 17 years
* Phase 1 PK expansion part in patients aged < 18 years to further assess PK/PD at the recommended phase 2 dose. In this part additional participants were enrolled to ensure that 6 patients in each of the 2 older age groups (2-6 and 7-17 years) were analyzed for PK before recruitment of infants < 2 years of age began.

In the phase 2 extension cohort (efficacy phase) of the study, eligible participants less than 18 years were enrolled according to a two-stage design and received blinatumomab at the recommended dose level (5/15 μg/m²/day).

The study consisted of a screening period, a treatment period, and an End of Core Study visit 30 days after last dose of study medication. A treatment cycle consisted of a continuous intravenous (cIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks. Participants who achieved complete remission (CR) within 2 cycles of treatment could receive up to 3 additional consolidation cycles of blinatumomab. Instead of consolidation cycles with blinatumomab, participants could be withdrawn from blinatumomab treatment to receive chemotherapy or allogeneic HSCT as early as the first cycle, at the discretion of the investigator.

After the last treatment cycle and End of Core Study visit, all participants were followed for efficacy and survival for up to 24 months after treatment start. Participants who suffered a hematological relapse of B-precursor ALL during their follow-up period (at least 3 months after completion of treatment) had the possibility for retreatment with blinatumomab.

ELIGIBILITY:
Inclusion Criteria:

* Morphologic evidence of B-precursor ALL with > 25% blasts in bone marrow (M3) at study enrolment
* Age less than 18 years at enrollment
* Relapsed/refractory disease:

  * Second or later bone marrow relapse,
  * Any marrow relapse after allogeneic hematopoietic stem cell transplantation (HSCT), or
  * Refractory to other treatments: Patients in first relapse must have failed to achieve a CR following full standard reinduction chemotherapy regimen of at least 4 weeks duration. Patients who have not achieved a first remission must have failed a full standard induction regimen
* Karnofsky performance status more than or equal to 50% for patients more than or equal to 16 years and Lansky Performance Status (LPS) of more than or equal to 50% for patients less than 16 years
* Organ function requirements: All patients must have adequate renal and liver functions

Exclusion Criteria:

* Active acute or extensive chronic graft-versus-host disease (GvHD)
* Immunosuppressive agents to prevent or treat GvHD within 2 weeks prior to blinatumomab treatment
* Evidence for current central nervous system (CNS) involvement by ALL (CNS 2, CNS 3) or testicular involvement by ALL
* History of relevant CNS pathology or current relevant CNS pathology
* History of autoimmune disease with potential CNS involvement or current autoimmune disease
* Any HSCT within 3 months prior to blinatumomab treatment
* Cancer chemotherapy within 2 weeks prior to blinatumomab treatment (except for intrathecal chemotherapy and/or low dose maintenance therapy such as vinca alkaloids, mercaptopurine, methotrexate, glucocorticoids)
* Chemotherapy related toxicities that haven't resolved to less than or equal to Grade 2
* Radiotherapy within 2 weeks prior to blinatumomab treatment
* Immunotherapy (e.g. rituximab, alemtuzumab) within 6 weeks prior to blinatumomab treatment
* Any investigational product within 4 weeks prior to study entry
* Previous treatment with blinatumomab
* Active severe infection, any other concurrent disease or medical condition that could be exacerbated by the treatment or would seriously complicate compliance with the protocol
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HbsAg positive) or hepatitis C virus (anti-HCV positive)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arend von Stackelberg, MD, Study Chair — Charite University, Berlin, Germany; Lia Gore, MD, Study Chair — Children's Hospital Denver, USA
Locations (30):
- United States (11):
  - Children's Hospital Denver, Aurora, Colorado
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Cancer Center/ Baylor, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- St. Anna Kinderspital, Vienna, Austria
- Hospital for Sick Children, Toronto, Ontario, Canada
- France (3):
  - (CHU Besancon) Hopital Saint-Jaques, Besançon
  - Hôpital de la Timone (Enfants), Marseille
  - Hopital Robert Debré (AP-HP), Paris
- Germany (10):
  - Charité Campus Virchow Klinikum, Otto-Heubner-Centrum (OHC) für Kinder- und Jugendmedizin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt/Main, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Klinikum der Universität München, Dr. von Haunersches Kinderspital, München
  - Universitätsklinik für Kinder- und Jugendmedizin Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Italy (3):
  - University of Milano-Bicocca, Hospital San Gerardo, Monza
  - Dipartimento della Donna e del Bambino, Padua
  - The Bambino Gesù Children's Hospital, Rome
- Erasmus MC, Sophia Children's Hospital, Rotterdam, Netherlands

REFERENCES:
- [Derived] von Stackelberg A, Locatelli F, Zugmaier G, Handgretinger R, Trippett TM, Rizzari C, Bader P, O'Brien MM, Brethon B, Bhojwani D, Schlegel PG, Borkhardt A, Rheingold SR, Cooper TM, Zwaan CM, Barnette P, Messina C, Michel G, DuBois SG, Hu K, Zhu M, Whitlock JA, Gore L. Phase I/Phase II Study of Blinatumomab in Pediatric Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia. J Clin Oncol. 2016 Dec 20;34(36):4381-4389. doi: 10.1200/JCO.2016.67.3301. Epub 2016 Oct 31. PMID 27998223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 26 centers in Germany, France, Italy, the Netherlands, the United Kingdom, and the United States of America. Results are reported for the primary analysis with a data cut-off date of 12 January 2015.
Pre-assignment Details: The Phase 1 part of the study comprised 2 parts:
  * a dose evaluation/escalation part in patients aged 2 to 17 years to define the recommended phase 2 dose of blinatumomab (4 arms),
  * a pharmacokinetic (PK) expansion part in patients less than 18 years.
  The Phase 2 efficacy part enrolled patients at the recommended dose determined in phase 1.
Groups:
- Phase 1: Blinatumomab 5 µg/m²/Day: Dose Evaluation/Escalation: Blinatumomab was administered as a continuous intravenous (cIV) infusion at a constant daily flow rate of 5 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Phase 1: Blinatumomab 15 µg/m²/Day: Dose Evaluation/Escalation: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 15 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Phase 1: Blinatumomab 30 µg/m²/Day: Dose Evaluation/Escalation: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 30 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Phase 1: Blinatumomab 15/30 µg/m²/Day: Dose Evaluation/Escalation: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 15 µg/m²/day for the first week of cycle 1 and then at 30 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 30 µg/m²/day for up to five cycles of treatment.
- Phase 1: Blinatumomab 5/15 µg/m²/Day: PK Expansion: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/day for the first week of cycle 1 and then at 15 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 15 µg/m²/day for up to five cycles of treatment.
- Phase 2: Blinatumomab 5/15 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/day for the first week of cycle 1 and then at 15 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 15 µg/m²/day for up to five cycles of treatment.
Period: Overall Study
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 5/15 µg/m²/Day | Phase 2: Blinatumomab 5/15 µg/m²/Day
Started | 5 | 7 | 5 | 6 | 26 | 44
Completed | 0 (Completed 5 cycles) | 1 (Completed 5 cycles) | 0 (Completed 5 cycles) | 1 (Completed 5 cycles) | 0 (Completed 5 cycles) | 3 (Completed 5 cycles)
Not Completed | 5 | 6 | 5 | 5 | 26 | 41
Not completed — Hematopoietic Stem Cell Transplantation | 2 | 2 | 1 | 0 | 5 | 3
Not completed — Lack of Efficacy | 1 | 2 | 1 | 1 | 5 | 18
Not completed — Adverse Event | 1 | 1 | 2 | 2 | 3 | 1
Not completed — Other | 0 | 0 | 1 | 1 | 6 | 5
Not completed — Change of Chemotherapy | 1 | 1 | 0 | 0 | 1 | 4
Not completed — Disease Relapse | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 3 | 8
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Blinatumomab 5 µg/m²/Day: Blinatumomab was administered as a continuous intravenous (cIV) infusion at a constant daily flow rate of 5 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Phase 1: Blinatumomab 15 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 15 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Phase 1: Blinatumomab 30 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 30 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Phase 1: Blinatumomab 15/30 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 15 µg/m²/day for the first week of cycle 1 and then at 30 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 30 µg/m²/day for up to five cycles of treatment.
- Phase 1: Blinatumomab 5/15 µg/m²/Day; Phase 2: Blinatumomab 5/15 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/day for the first week of cycle 1 and then at 15 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 15 µg/m²/day for up to five cycles of treatment.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 5/15 µg/m²/Day | Phase 2: Blinatumomab 5/15 µg/m²/Day | Total
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 26 | 44 | 93
Age, Customized [Number; unit: participants]
  < 2 years | 0 | 0 | 0 | 0 | 8 | 2 | 10
  2 - 6 years | 3 | 5 | 2 | 4 | 9 | 11 | 34
  7 - 17 years | 2 | 2 | 3 | 2 | 9 | 31 | 49
Gender [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 1 | 11 | 12 | 33
  Male | 2 | 3 | 3 | 5 | 15 | 32 | 60
Race/Ethnicity, Customized [Number; unit: participants] — Race was not recorded for any patient from France and for two further patients.
  participants
    White | 5 | 7 | 5 | 5 | 22 | 33 | 77
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    American Indian or Alaska native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or other Pacific islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Other | 0 | 0 | 0 | 1 | 3 | 5 | 9
    Unknown | 0 | 0 | 0 | 0 | 1 | 6 | 7
Prior Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) [Number; unit: participants]
  Yes | 3 | 6 | 2 | 4 | 15 | 25 | 55
  No | 2 | 1 | 3 | 2 | 11 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: The maximum tolerated dose (MTD) was defined as one or fewer out of 6 participants experiencing a dose limiting toxicity (DLT) or the maximum administered dose (MAD).
  A dose limiting toxicity is any Grade ≥ 3 adverse event related to study drug, Grade 3 fatigue, headache, insomnia, fever, hypotension or infection were not considered dose limiting toxicities. Laboratory parameters of Grade ≥ 3 but not considered as clinically relevant and/or responding to routine medical management, thrombocytopenia, leukopenia (including neutropenia and lymphopenia), and anemia were not considered dose limiting toxicities.
Time Frame: Cycle 1, 28 days
Population: Participants in the Phase 1 dose evaluation/escalation part of the study
Measure: Number; unit: participants
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day
Number analyzed (Participants) | 5 | 7 | 5 | 6
participants | 0 | 1 | 2 | 1

2. Primary Outcome: Percentage of Participants With Complete Remission in the First Two Cycles
Description: Hematological assessments were performed from bone marrow biopsy samples. All hematological assessments of bone marrow were reviewed in a central laboratory. Complete remission (CR) was defined as
  * M1 bone marrow (bone marrow blasts < 5%)
  * No evidence of circulating blasts or extra-medullary disease
  Complete remission includes participants with incomplete recovery of peripheral blood counts.
Time Frame: Cycles 1 and 2 (12 weeks)
Population: The full analysis set includes all participants who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1+2: Blinatumomab 5/15 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/ day for the first week of cycle 1 and then at 15 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 15 µg/m²/day for up to five cycles of treatment.
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 5/15 µg/m²/Day | Phase 2: Blinatumomab 5/15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 26 | 44 | 70
percentage of participants | 20.0 [0.5 to 71.6] | 42.9 [9.9 to 81.6] | 20.0 [0.5 to 71.6] | 33.3 [4.3 to 77.7] | 50.0 [29.9 to 70.1] | 31.8 [18.6 to 47.6] | 38.6 [27.2 to 51.0]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity (or intensity) of adverse events (AEs) was assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), v4.03 and according to the following:
  Grade 1 - Mild adverse event; Grade 2 - Moderate adverse event; Grade 3 - Severe and undesirable adverse event; Grade 4 - Life-threatening or disabling adverse event; Grade 5 - Death. The investigator used medical judgment to determine if there was a causal relationship (ie, related, unrelated) between an adverse event and blinatumomab.
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion in the core study or from the start of the first retreatment cycle infusion to 30 days after the end of the last retreatment cycle, median treatment duration was 28 days
Population: Full analysis set
Measure: Number; unit: participants
Groups:
- Phase 1+2: Blinatumomab 5/15 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/day for the first week of cycle 1 and then at 15 µg/m²/day for 3 weeks followed by a treatment-free interval of 2 weeks. Participants received subsequent cycles at 15 µg/m²/day for up to five cycles of treatment.
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day
Number analyzed (Participants) | 5 | 7 | 70 | 6 | 5
participants
  Any adverse event (AE) | 5 | 7 | 70 | 6 | 5
  Adverse event of at least CTC grade 3 | 4 | 7 | 61 | 6 | 5
  Serious adverse event (SAEs) | 4 | 4 | 39 | 4 | 3
  SAE of at least grade 3 | 4 | 3 | 28 | 4 | 3
  AE leading to interruption of study drug | 0 | 0 | 10 | 2 | 2
  AE leading to discontinuation of study drug | 1 | 1 | 4 | 2 | 2
  Adverse event leading to death | 0 | 1 | 8 | 3 | 1
  Treatment-related adverse event (TRAE) | 5 | 6 | 59 | 5 | 5
  TRAE of at least CTC grade 3 | 4 | 5 | 38 | 4 | 5
  Treatment-related serious adverse event | 3 | 2 | 15 | 1 | 2
  TRAE leading to discontinuation of study drug | 1 | 1 | 2 | 1 | 2
  TRAE leading to death | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Steady State Concentration of Blinatumomab
Description: Blinatumomab serum concentrations were quantified in all patients during the first 2 treatment cycles in the phase 1 part of the study only. Blinatumomab concentrations were quantified using a validated bioassay, the lower limit of quantification was 50 pg/mL. Steady state serum concentration (Css) was presumed on day 1, approximately 5 half-lives after the start of the IV infusion.
  The steady state serum concentration reported is the mean of the observed concentrations collected after during cycles 1 and 2.
Time Frame: Cycles 1 and 2 during the IV infusion on day 3 (at least 48 hours after start of infusion) and days 8, 15 and 22 (steady state) and day 29 at End of Infusion (EoI) and 2, 4, and 8 hours after EoI for ages ≥ 2 years.
Population: Phase 1 participants with available blinatumomab concentration data
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Phase 1: Blinatumomab 5 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/day.
- Phase 1: Blinatumomab 15 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 15 µg/m²/day.
- Phase 1: Blinatumomab 30 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 30 µg/m²/day.
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day
Number analyzed (Participants) | 27 | 34 | 7
pg/mL
  Cycle 1 (N = 27, 34, 7) | 162 (179) | 533 (392) | 1520 (1020)
  Cycle 2 (N = 3, 13, 5) | 456 (288) | 866 (655) | 1150 (701)

5. Secondary Outcome: Time to Hematological Relapse (Duration of Response)
Description: Time to hematological relapse was measured only for participants in remission and was measured from the time the participant first achieved remission until first documented relapse or death due to disease progression. Participants without a documented relapse (hematological or extramedullary) and who did not die were censored at the time of their last bone marrow assessment or their last survival follow-up visit confirming remission. Participants who died without having reported hematological relapse or without showing any clinical sign of disease progression were censored on their date of death.
  Hematological relapse is defined as the proportion of blasts in bone marrow > 25% following documented remission, or extramedullary relapse.
  Time to hematological relapse was analyzed by Kaplan-Meier methods and the median observation time was calculated by the reverse Kaplan Meier method.
Time Frame: Up to the data cut-off date of 12 January 2015; median observation time was 23.5 months for phase 1 and 11.5 months for phase 2.
Population: Full analysis set with complete remission
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1: Blinatumomab: Blinatumomab was administered as a continuous intravenous (cIV) infusion at a constant daily flow rate ranging from 5 to 30 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
Arm/Group | Phase 1: Blinatumomab | Phase 2: Blinatumomab 5/15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day
Number analyzed (Participants) | 21 | 14 | 27
months | 10.3 [3.9 to 16.4] | 3.4 [1.7 to NA] — Could not be estimated due to the low number of events | 5.2 [2.3 to 16.4]

6. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was measured for all participants from the first treatment of blinatumomab until death due to any cause or the date of the last follow-up. Participants who did not die were censored on the last documented visit date or the date of the last contact when the patient was last known to have been alive. For patients who withdrew their informed consent only information until the date of withdrawal was analyzed.
  Overall survival was estimated using Kaplan-Meier methods. The median follow-up time with respect to overall survival was calculated by the reverse Kaplan-Meier method.
Time Frame: Up to the data cut-off date of 12 January 2015; median observation time was 23.5 months for phase 1 and 11.6 months for phase 2.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Blinatumomab | Phase 2: Blinatumomab 5/15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day
Number analyzed (Participants) | 49 | 44 | 70
months | 6.5 [3.6 to 10.6] | 8.2 [4.0 to 14.6] | 7.5 [4.0 to 11.8]

7. Secondary Outcome: Relapse-free Survival
Description: Relapse-free survival (RFS) was assessed for participants who achieved a complete remission during the core study and was measured from the time the participant first achieved remission until first documented relapse or death due to any cause. Participants without a documented relapse (hematological or extramedullary) or who did not die were censored at the time of their last bone marrow assessment or their last survival follow-up visit confirming remission.
  Relapse free survival was estimated using Kaplan-Meier methods and the median observation time was calculated by the reverse Kaplan-Meier method.
Time Frame: as for outcome 5
Population: Full analysis set with complete remission
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1: Blinatumomab: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate ranging from 5 to 30 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
Arm/Group | Phase 1: Blinatumomab | Phase 2: Blinatumomab 5/15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day
Number analyzed (Participants) | 21 | 14 | 27
months | 7.9 [3.0 to 12.4] | 3.4 [1.7 to 13.9] | 4.4 [2.3 to 12.1]

8. Secondary Outcome: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant During Blinatumomab Induced Remission
Description: The percentage of participants who received allogeneic hematopoietic stem cell transplantation (HSCT) while in remission due to treatment with blinatumomab during the first two cycles, and received no further anti-leukemic medication before HSCT.
Time Frame: Up to the data cut-off date of 12 January 2015; Maximum duration on study was 24 months in phase 1 and 15 months for phase 2.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 5/15 µg/m²/Day | Phase 2: Blinatumomab 5/15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 26 | 44 | 70
percentage of participants | 20.0 [0.5 to 71.6] | 28.6 [3.7 to 71.0] | 20.0 [0.5 to 71.6] | 16.7 [0.4 to 64.1] | 30.8 [14.3 to 51.8] | 11.4 [3.8 to 24.6] | 18.6 [10.3 to 29.7]

9. Secondary Outcome: Number of Participants Who Developed Anti-blinatumomab Antibodies
Description: Antibodies to blinatumomab were detected using an electrochemiluminescence (ECL)-based assay.
Time Frame: Predose up until 30 days after last dose of study medication; median treatment duration was 28 days.
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 5/15 µg/m²/Day | Phase 2: Blinatumomab 5/15 µg/m²/Day
Number analyzed (Participants) | 5 | 7 | 5 | 6 | 26 | 44
participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Serum Cytokine Peak Levels
Description: The activation of immune effector cells was monitored by the measurement of peripheral blood cytokine levels including interleukin (IL)-2, IL-4, IL-6, IL-10, tumor necrosis factor-alpha (TNF-α) and interferon gamma (IFN-ɣ) using cytometric bead assays. The limit of detection of the assay (LOD) was 20 pg/mL and the lower limit of quantification (LLOQ) was 125 pg/mL. Data below LOD were set to 10 pg/mL while data < LOQ and > LOD were reported as measured.
Time Frame: Cycle 1 and 2 day 1 (prior to infusion, 2 and 6 hours after infusion start), day 2 and day 3.
Population: Phase 1 full analysis set participants with available data
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day
Number analyzed (Participants) | 31 | 14 | 5
pg/mL
  IL-6: Cycle 1 Week 1 (N=31, 13, 5) | 4970 (17000) | 1780 (2620) | 23400 (24100)
  IL-6: Cycle 2 Week 1 (N=4, 14, 5) | 526 (844) | 892 (2370) | 40.4 (68.0)
  IL-10: Cycle 1 Week 1 (N=31, 13, 5) | 562 (710) | 1400 (2030) | 3170 (1720)
  IL-10: Cycle 2 Week 1 (N=4, 14, 5) | 519 (497) | 432 (692) | 277 (308)
  IFN-ɣ: Cycle 1 Week 1 (N=31, 13, 5) | 207 (516) | 539 (1240) | 2260 (1540)
  IFN-ɣ: Cycle 2 Week 1 (N=4, 14, 5) | 51.8 (65.6) | 47.6 (51.5) | 22.8 (28.6)
  IL-2: Cycle 1 Week 1 (N=31, 13, 5) | 22.7 (23) | 93.9 (150) | 900 (1390)
  IL-2: Cycle 2 Week 1 (N=4, 14, 5) | 10.0 (0.00) | 14.3 (8.84) | 10.0 (0.00)
  TNF-α: Cycle 1 Week 1 (N=31, 13, 5) | 87.3 (241) | 60.2 (127) | 285 (306)
  TNF-α: Cycle 2 Week 1 (N=4, 14, 5) | 10.0 (0.00) | 10.0 (0.00) | 10.0 (0.00)
  IL-4: Cycle 1 Week 1 (N=0, 0, 0) | NA (NA) — Serum IL-4 levels were below detection limit (< 20 pg/mL) in all participants studied. | NA (NA) — Serum IL-4 levels were below detection limit (< 20 pg/mL) in all participants studied. | NA (NA) — Serum IL-4 levels were below detection limit (< 20 pg/mL) in all participants studied.
  IL-4: Cycle 2 Week 1 (N=0, 0, 0) | NA (NA) — Serum IL-4 levels were below detection limit (< 20 pg/mL) in all participants studied. | NA (NA) — Serum IL-4 levels were below detection limit (< 20 pg/mL) in all participants studied. | NA (NA) — Serum IL-4 levels were below detection limit (< 20 pg/mL) in all participants studied.

ADVERSE EVENTS:
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion in the core study or from the start of the first retreatment cycle infusion to 30 days after the end of the last retreatment cycle, median treatment duration was 28 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Phase 1: Blinatumomab 5 µg/m²/Day: Blinatumomab was administered as a continuous intravenous infusion at a constant daily flow rate of 5 µg/m²/day over 4 weeks followed by a treatment-free interval of 2 weeks for up to five cycles of treatment.
- Total: All Participants who received blinatumomab administered as a continuous intravenous infusion at a constant daily flow rate.
Arm/Group | Phase 1: Blinatumomab 5 µg/m²/Day | Phase 1: Blinatumomab 15 µg/m²/Day | Phase 1+2: Blinatumomab 5/15 µg/m²/Day | Phase 1: Blinatumomab 15/30 µg/m²/Day | Phase 1: Blinatumomab 30 µg/m²/Day | Total
Serious Adverse Events (participants affected / at risk) | 4/5 | 4/7 | 39/70 | 4/6 | 3/5 | 54/93
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 70/70 | 6/6 | 5/5 | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Blinatumomab 5 µg/m²/Day (N=5) | Phase 1: Blinatumomab 15 µg/m²/Day (N=7) | Phase 1+2: Blinatumomab 5/15 µg/m²/Day (N=70) | Phase 1: Blinatumomab 15/30 µg/m²/Day (N=6) | Phase 1: Blinatumomab 30 µg/m²/Day (N=5) | Total (N=93)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 0 | 0 | 8
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 1 | 0 | 2
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 2 | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 1 | 8 | 0 | 0 | 11
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 4 | 0 | 2 | 7
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 3
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Enterococcus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Escherichia test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Stenotrophomonas test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Atonic seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 3
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1 | 1 | 6
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Blinatumomab 5 µg/m²/Day (N=5) | Phase 1: Blinatumomab 15 µg/m²/Day (N=7) | Phase 1+2: Blinatumomab 5/15 µg/m²/Day (N=70) | Phase 1: Blinatumomab 15/30 µg/m²/Day (N=6) | Phase 1: Blinatumomab 30 µg/m²/Day (N=5) | Total (N=93)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 29 | 2 | 4 | 40
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2 | 3 | 1 | 1 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 1 | 0 | 9
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 9 | 1 | 2 | 14
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 12 | 0 | 0 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 14 | 1 | 2 | 21
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 3 | 1 | 2 | 6
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 5 | 1 | 1 | 7
Tachycardia (Cardiac disorders) | 0 | 0 | 3 | 0 | 1 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 2 | 0 | 1 | 3
Eyelid haematoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 2 | 0 | 0 | 3
Ocular icterus (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 2
Photophobia (Eye disorders) | 0 | 1 | 2 | 0 | 1 | 4
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 13 | 0 | 1 | 20
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 6 | 2 | 0 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 9 | 0 | 1 | 14
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 3
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 23 | 1 | 1 | 28
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2 | 17 | 2 | 2 | 25
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Application site scab (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 2 | 0 | 0 | 3
Chills (General disorders) | 0 | 0 | 3 | 0 | 1 | 4
Face oedema (General disorders) | 1 | 0 | 1 | 0 | 1 | 3
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 5 | 0 | 2 | 11
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 4 | 0 | 0 | 4
Oedema (General disorders) | 0 | 0 | 3 | 2 | 0 | 5
Oedema peripheral (General disorders) | 1 | 0 | 5 | 0 | 1 | 7
Pain (General disorders) | 1 | 2 | 6 | 3 | 0 | 12
Pyrexia (General disorders) | 4 | 7 | 54 | 4 | 5 | 74
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 2
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 4 | 2 | 2 | 9
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 2
Adenovirus infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2
BK virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 4
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Legionella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 7 | 0 | 0 | 7
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Viral myositis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 3
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 4 | 0 | 0 | 5
Alanine aminotransferase increased (Investigations) | 1 | 0 | 13 | 2 | 2 | 18
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 10 | 2 | 2 | 16
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 4 | 1 | 3 | 9
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0 | 2 | 4
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Blood fibrinogen increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood immunoglobulin A decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 4 | 1 | 0 | 0 | 5
Blood immunoglobulin M decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 7 | 0 | 2 | 10
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1 | 1 | 0 | 0 | 2
Electroencephalogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 2 | 6 | 1 | 1 | 10
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 2 | 3 | 2 | 0 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 3 | 1 | 1 | 5
Neutrophil count decreased (Investigations) | 0 | 0 | 9 | 3 | 2 | 14
Platelet count decreased (Investigations) | 0 | 0 | 10 | 2 | 1 | 13
Protein total decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 3
Roseolovirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 4 | 1 | 0 | 5
Weight increased (Investigations) | 0 | 1 | 12 | 2 | 1 | 16
White blood cell count decreased (Investigations) | 0 | 0 | 8 | 3 | 2 | 13
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 1 | 0 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 2 | 0 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 8 | 1 | 1 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 15 | 3 | 0 | 22
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 1 | 0 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 2 | 0 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 10 | 2 | 0 | 12
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 14 | 0 | 2 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7 | 0 | 1 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 8 | 2 | 2 | 17
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0 | 0 | 5
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 4 | 20 | 0 | 2 | 31
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 4 | 2 | 0 | 7
Agitation (Psychiatric disorders) | 0 | 1 | 3 | 0 | 1 | 5
Anxiety (Psychiatric disorders) | 1 | 0 | 4 | 0 | 1 | 6
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 3
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 3
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 3
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Renal tubular disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 13 | 0 | 2 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 10 | 1 | 0 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 3
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 1 | 7
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Infusion (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 1
Oxygen supplementation (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0 | 2
Parenteral nutrition (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 2 | 2 | 0 | 4
Flushing (Vascular disorders) | 0 | 0 | 3 | 0 | 1 | 4
Haematoma (Vascular disorders) | 0 | 0 | 2 | 0 | 1 | 3
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 5 | 18 | 2 | 1 | 26
Hypotension (Vascular disorders) | 0 | 1 | 10 | 2 | 1 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.